CLINICAL TRIAL: NCT01619943
Title: Prediction Value of the Canadian CT Head Rule and the New Orleans Criteria for Positive Head CT Scan and Acute Neurosurgical Procedures in Minor Head Trauma: a Multicenter External Validation Study
Brief Title: The Value of the Canadian CT Head Rule and the New Orleans Criteria in Minor Head Trauma
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nouira, Professor, University of Monastir
Other Study IDs: Head injury
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Minor Head Injury
Keywords: Minor head injury; CT scan; Canadian CT Head Rules; The New Orleans Criteria
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with minor head injury: MHI is defined as a blunt trauma to the head within 24 hours with a Glasgow Coma Scale (GCS) score of 13 to 15 and at least one of the following: history of loss of consciousness, short-term memory deficit, amnesia for the traumatic event, post-traumatic seizure, vomiting, headache, external evidence of injury above the clavicles, confusion, and neurologic deficit.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — clinical follow up
  Other Names: clinical follow up
Other: no intervention — no intervention

SUMMARY:
The New Orleans Criteria (NOC) and the Canadian CT Head Rules (CCHR) have been developed to decrease the number of normal computed tomography (CT) in mild head injury (MHI). The aim is to compare the clinical performance of these 2 decision rules for indentifying patients with intracranial traumatic lesions and those who required an emergent neurosurgical intervention following MHI.

DETAILED DESCRIPTION:
A multicenter external validation study in 7 Tunisian teaching and non teaching hospitals including patients with MHI defined as a blunt trauma to the head within 24 hours with a Glasgow Coma Scale (GCS) score of 13 to 15 and at least one of the following: history of loss of consciousness, short-term memory deficit, amnesia for the traumatic event, post-traumatic seizure, vomiting, headache, external evidence of injury above the clavicles, confusion, and neurologic deficit. Primary outcome was need for neurosurgical intervention defined as either death or craniotomy, or the need of endotracheal intubation within 30 days of the traumatic event. Secondary outcome was the presence of traumatic lesions on head CT scan. Comparaision of both decision rules using sensitivity specifications, positive and negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute MHI was defined as a patient having a blunt trauma to the head within 24 hours with a Glasgow Coma Scale (GCS) of 13 to 15 and at least 1 of the following risk factors: history of loss of consciousness, short-term memory deficit, amnesia for the traumatic event, post-traumatic seizure, vomiting, headache, external evidence of injury above the clavicles, confusion, and neurologic deficit.

Exclusion Criteria:

* Patients are excluded from the study if they are younger than 10 years, had GCS score of less than 13 or instable vital signs, came to the ED more than 24 hours after head trauma, were pregnant, were taking warfarin or had bleeding disorder, had an obvious penetrating skull injury or had contraindications for CT.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MHI defined as a blunt trauma to the head within 24 hours with a Glasgow Coma Scale (GCS) score of 13 to 15 and at least one of the following: history of loss of consciousness, short-term memory deficit, amnesia for the traumatic event, post-traumatic seizure, vomiting, headache, external evidence of injury above the clavicles, confusion, and neurologic deficit.
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Prof, Principal Investigator — Monastir Hospital
Locations (3):
- Tunisia (3):
  - University hospital of Monastir, Monastir, Monastir Governorate
  - University Hospital of Monastir, Monastir, Monstir
  - Fattouma Bourguiba University Hospital, Monastir